CLINICAL TRIAL: NCT01007708
Title: The Safety and Efficacy of Topical IDP-108 Versus Vehicle in Patients With Onychomycosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPSI-IDP-108-P3-02
Record Dates: First submitted 2009-11-03; First posted 2009-11-04 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDP-108 (Experimental)
  Interventions: Drug: IDP-108
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: IDP-108 — Topical application once a day for 48 weeks
  Arms: IDP-108
Drug: Vehicle — Topical application once a day for 48 weeks
  Arms: Vehicle

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of topical application of IDP-108 versus vehicle in treating patients with onychomycosis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed onychomycosis of the target nail
* Presence of mild to moderate onychomycosis, defined as 20 - 50% of the area of the target nail being clinically affected
* Has a positive KOH examination from the target nail
* Has a positive dermatophyte culture from the target nail

Exclusion Criteria:

* Presence of any disease or condition that might cause nail abnormalities or may interfere with the evaluation of the study drug
* Use of any systemic antifungal therapy within 4 weeks prior to the Screening visit or non-responsive to systemic antifungal therapy for onychomycosis
* Use of any prescription or over-the-counter topical antifungal therapy for the toenails within 4 weeks prior to the Screening visit
* Woman who is pregnant, nursing an infant, or planning a pregnancy during the study period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who achieve clinical cure | 52 weeks

SECONDARY OUTCOMES:
Percentage of patients who achieve clinical efficacy | 52 weeks
Percentage of patients who achieve mycologic cure | 52 weeks

CONTACTS AND LOCATIONS:
Locations (44):
- United States (36):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Impact Clinical Trials, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Specialists, Inc., Oceanside, California
  - Skin Surgery Medical Group, Inc., San Diego, California
  - Center for Clinical Research, San Francisco, California
  - Radiant Research, Santa Rosa, California
  - Colorado Medical Research Center Inc, Denver, Colorado
  - Ameriderm Research, Jacksonville, Florida
  - FXM Research Corp., Miami, Florida
  - MedaPhase Inc., Newnan, Georgia
  - Northwest Clinical Trials Nampa, Nampa, Idaho
  - DuPage Medical Group, Naperville, Illinois
  - Deaconess Clinic, Inc., Evansville, Indiana
  - South Bend Clinic, South Bend, Indiana
  - David Fivenson, MD, Dermatology, PLLC, Ann Arbor, Michigan
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - The Dermatology Group, P.C., Verona, New Jersey
  - Fran E. Cook-Bolden, MD, New York, New York
  - Skin Search of Rochester, Inc, Rochester, New York
  - DermResearchCenter of New York, Inc., Stony Brook, New York
  - University of North Carolina Hospitals and School of Medicine, Chapel Hill, North Carolina
  - New Hanover Medical Research, Wilmington, North Carolina
  - Brodell Medical, Inc, Warren, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Oregon Medical Center, PC, Portland, Oregon
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Dermatology East, Germantown, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc., Austin, Texas
  - Modern Research Associates, PLLC, Dallas, Texas
  - Suzanne Bruce and Associates, PA The Center for Skin Research, Houston, Texas
  - Endeavor Clinical Trials, PA, San Antonio, Texas
  - Premier Clinical Research, Spokane, Washington
  - Madison Skin & Research, Inc., Madison, Wisconsin
- Canada (8):
  - Guildford Dermatology Specialists, Surrey, British Columbia
  - Dermadvances Research, Winnipeg, Manitoba
  - NewLab Clinical Research, St. John's, Newfoundland and Labrador
  - Lynderm Research, Inc., Markham, Ontario
  - The Centre for Dermatology & Cosmetic Surgery, Richmond Hill, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Windsor Clinical Research, Windsor, Ontario
  - Beatrice Wang, MD, Westmount, Quebec

REFERENCES:
- [Derived] Gupta AK, Elewski BE, Sugarman JL, Ieda C, Kawabata H, Kang R, Pillai R, Olin JT, Watanabe S. The efficacy and safety of efinaconazole 10% solution for treatment of mild to moderate onychomycosis: a pooled analysis of two phase 3 randomized trials. J Drugs Dermatol. 2014 Jul;13(7):815-20. PMID 25007364